CLINICAL TRIAL: NCT05566886
Title: Multi Parameter Vital Signs Monitoring by the Corsano CardioWatch 287-2 Validation Study
Brief Title: Validation of a Vital Signs Monitoring Wristband
Acronym: MULTI-VITAL
Status: Completed | Type: Observational
Sponsor: Corsano Health B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: MULTI-VITAL
Record Dates: First submitted 2022-09-20; First posted 2022-10-04 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease
Keywords: Vital signs; Blood pressure; Oxygen saturation; Heart rate; Respiratory rate
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Continuous measurement of photoplethysmography at the wrist — Patients receive a wristband that uses multi-color LEDs to measure pulsations at the wrist.

SUMMARY:
Today, continuous monitoring of vital signs remains a challenge since it generally requires the patient to be connected to multiple wired sensors, which restricts patient mobility in the intra-mural setting and complicates home monitoring in the extra-mural setting. Wearable devices on the wrist, although emerging, are often not clinically validated or limited to the monitoring of one or two vital signs.

This study aims to validate the Corsano CardioWatch 287-2 for the continuous monitoring of heart rate at ≤ 4 bpm root mean squared error (RMSE); interbeat intervals at ≤ 50 ms RMSE; breathing rate at ≤ 2 brpm RMSE; and peripheral oxygen saturation at ≤ 3 percentage point RMSE. Also, this study aims to validate the Corsano CardioWatch 287-2 for the measurement of non-invasive blood pressure according to ISO 81060-2:2018.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old;
* undergoing invasive monitoring, like coronary angiography;
* able to provide consent.

Exclusion Criteria:

Patients

* who cannot wear the Corsano CardioWatch 287 due to reasons such as allergic reactions, wounds, amputations etc.;
* unable or not willing to sign informed consent;
* with significant mental or cognitive impairment;
* who do not have a suitable entry site for the invasive arterial line
* who do not comply to criteria established by ISO 81060-2:2018.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Reinier de Graaf Gasthuis, Delft, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monnink SHJ, van Vliet M, Kuiper MJ, Constandse JC, Hoftijzer D, Muller M, Ronner E. Clinical evaluation of a smart wristband for monitoring oxygen saturation, pulse rate, and respiratory rate. J Clin Monit Comput. 2025 Apr;39(2):451-457. doi: 10.1007/s10877-024-01229-z. Epub 2024 Oct 10. PMID 39388061
- [Derived] van Vliet M, Monnink SHJ, Kuiper MJ, Constandse JC, Hoftijzer D, Ronner E. Evaluation of a novel cuffless photoplethysmography-based wristband for measuring blood pressure according to the regulatory standards. Eur Heart J Digit Health. 2024 Feb 8;5(3):335-343. doi: 10.1093/ehjdh/ztae006. eCollection 2024 May. PMID 38774367

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 124 subjects undergoing heart catheterization were screened. 24 participants were not included due to:
  * Lateral difference exceeding limits (n=8)
  * Arm circumference not within range (n=1)
  * Atrial fibrillation or arrhythmia (n=5)
  * Peripheral artery disease (n=3)
  * Unforeseen difficulties during procedure (n=2)
  * Other medical reasons (e.g., isolation for infection) (n=1)
  * Technical difficulties (measurement not started) (n=1)
  * Procedure canceled or postponed (n=3)
Groups:
- Main Study Group: Subjects undergoing heart catheterization as standard of care.
Period: Overall Study
Arm/Group | Main Study Group
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Main Study Group
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 67
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Skin colour (Fitzpatrick) [Count of Participants; unit: Participants]
  Fitzpatrick Class I-II | 81
  Fitzpatrick Class III-IV | 16
  Fitzpatrick Class V-VI | 3

OUTCOME MEASURES:

1. Primary Outcome: RMSE of Heart Rate
Description: Root-mean-squared error between PPG measured and gold standard measured heart rate
Time Frame: 30 minutes
Measure: Mean (Full Range); unit: beats per minute
Units Other Than Participants: epochs (28 second)
Arm/Group | Main Study Group
Number analyzed (Participants) | 100
Number analyzed (epochs (28 second)) | 945
beats per minute | 1.3 [-5.5 to 4.2]

2. Primary Outcome: RMSE of Respiratory Rate
Description: Root-mean-squared error between PPG measured and gold standard measured respiratory rate
Time Frame: 30 minutes
Measure: Mean (Full Range); unit: breaths per minute
Units Other Than Participants: epochs (28 second)
Arm/Group | Main Study Group
Number analyzed (Participants) | 100
Number analyzed (epochs (28 second)) | 945
breaths per minute | 0.9 [-2.1 to 2]

3. Primary Outcome: RMSE of Oxygen Saturation
Description: Root-mean-squared error between PPG measured and gold standard measured oxygen saturation
Time Frame: 30 minutes
Measure: Mean (Full Range); unit: % of SpO2
Units Other Than Participants: epochs (28 second)
Arm/Group | Main Study Group
Number analyzed (Participants) | 100
Number analyzed (epochs (28 second)) | 945
% of SpO2 | 1.6 [-3.2 to 3.9]

4. Primary Outcome: RMSE of Blood Pressure
Description: Root-mean-squared error between PPG measured and gold standard measured blood pressure (systolic blood pressure and diastolic blood pressure)
Time Frame: 30 minutes
Population: 100 subjects were included, however, 3 individuals did not meet pre-specified dampening criteria
  As a result data of 97 patients and 420 measurement pairs was included in the analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: paired samples
Groups:
- Main Study Group: Subjects undergoing heart catheterization as standard of care. 3 individuals did not meet pre-specified dampening criteria
Arm/Group | Main Study Group
Number analyzed (Participants) | 97
Number analyzed (paired samples) | 420
mmHg
  Systolic Blood Pressure | 3.7 (4.4)
  Diastolic Blood Pressure | 2.5 (3.7)

ADVERSE EVENTS:
Time Frame: During study intervention alone (during 1 hour study duration)
Arm/Group | Main Study Group
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-04): https://cdn.clinicaltrials.gov/large-docs/86/NCT05566886/Prot_SAP_000.pdf